CLINICAL TRIAL: NCT03552705
Title: Novel Strategies to Combat Post-Traumatic Osteoarthritis (PTOA):The Effects of Tranexamic Acid on Joint Inflammation and Cartilage Health in Anterior Cruciate Ligament Injured Patients
Brief Title: The Effects of Tranexamic Acid on Joint Inflammation and Cartilage Health in Anterior Cruciate Ligament Injured Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Constance R. Chu, MD, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 46092; CDMRP-PR171647 (Other Grant/Funding Number: DoD)
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Anterior Cruciate Ligament Reconstruction
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic Acid (Experimental): 5-day course of standard adult oral tranexamic acid dosage of 1300 mg taken 3 times a day (3900 mg/day) and intravenous tranexamic acid during ACL reconstruction surgery (1 gram of iv TXA just prior to incision and 1 gram of iv TXA just prior to wound closure)
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): 5-day course of placebo and intravenous saline during ACL reconstruction surgery
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Tranexamic Acid — 5-day course of oral standard adult oral tranexamic acid dosage of 1300 mg taken 3 times a day (3900 mg/day) and intravenous tranexamic acid during ACL reconstruction surgery (1 gram of iv TXA just prior to incision and 1 gram of iv TXA just prior to wound closure)
  Arms: Tranexamic Acid
Drug: Placebos — 5-day course of oral placebo and intravenous saline during ACL reconstruction surgery
  Arms: Placebo

SUMMARY:
Patients who tear their ACL are at high risk for developing arthritis (post-traumatic osteoarthritis-PTOA) just 10 years later. Joint bleeding and inflammation contribute to deterioration of joint health. This study will determine whether treatment with Tranexamic Acid (TXA), an FDA approved medication that reduces bleeding right after ACL injury and reconstructive surgery reduces inflammation and improves joint health as a new strategy to prevent or delay the onset of PTOA.

ELIGIBILITY:
Inclusion Criteria:

* age 18-30 years
* within 4 days of unilateral ACL injury
* presence of effusion/hemarthrosis.

Exclusion Criteria:

* inflammatory arthritis, radiographic osteoarthritis (K-L Grade 2 or higher), gout/ pseudogout
* systemic or acute illness requiring medications
* concomitant knee injury aside from meniscus tear and MCL tear not requiring surgery
* prior surgery to either knee
* prior injury to either knee requiring crutches
* history of thromboembolic disease
* current use of combination hormonal contraception
* chronic NSAID use
* cortisone injection to either knee within the prior 3 months
* not indicated for or unable to undergo ACLR within 3 months of injury

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2026-01-14 (Estimated); Study Completion 2026-01-14 (Estimated)

PRIMARY OUTCOMES:
Synovial fluid IL-1 | Day 5
  To determine whether TXA administered acutely after ACL injury reduces synovial fluid markers of inflammation and cartilage degradation
Patient-Reported Outcomes (PRO): Knee injury and Osteoarthritis Outcome Score (KOOS) | 6 months post-ACLR
  To determine whether TXA administered acutely after ACL injury and during ACLR surgery improves PRO (KOOS Quality of Life) at 6 months after ACLR. The Knee injury and Osteoarthritis Outcome Score (KOOS) assesses a patient's opinion about their knee and associated problems. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated.

SECONDARY OUTCOMES:
Quantitative MRI (qMRI) | 6 months post-ACLR
  To determine whether TXA administered acutely after ACL injury and during ACLR surgery improves cartilage subsurface matrix structure assessed by qMRI UTE-T2* at 6 months after ACLR
Quantitative MRI | 2 years post-ACLR
  To determine whether TXA administered acutely after ACL injury and during ACLR surgery improves cartilage subsurface matrix structure assessed by qMRI UTE-T2* at 2 years after ACLR
Patient-Reported Outcomes (PRO): Knee injury and Osteoarthritis Outcome Score (KOOS) | 2 years post-ACLR
  To determine whether TXA administered acutely after ACL injury and during ACLR surgery improves PRO (KOOS Quality of Life) at 2 years after ACLR. The Knee injury and Osteoarthritis Outcome Score (KOOS) assesses a patient's opinion about their knee and associated problems. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Constance Chu, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States